CLINICAL TRIAL: NCT06152640
Title: A New Neuroregulatory Technology for the Therapy of AN Based on the Pathological Neural Network of ACC: A Multicenter Randomized Controlled Study
Brief Title: A New Neuroregulatory Technology for the Therapy of AN Based on the Pathological Neural Network of ACC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Huadong Hospital (Other); Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jue CHEN, Director of Psychosomatic Department in Shanghai Mental Health Center, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHDC12023122
Record Dates: First submitted 2023-11-16; First posted 2023-12-01 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Feeding and Eating Disorders
Keywords: anorexia nervosa; Deep transcranial magnetic stimulation; anterior cingulate cortex
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dTMS treatment group (Experimental): dTMS treatment group has 40 patients with dTMS intervention using real coils, targeting ACC, given once per day, for 28 days, with a total of 28 treatments.
  Interventions: Device: Deep transcranial magnetic stimulation; Other: Basic treatment
- pseudo-stimulation group (Sham Comparator): Pseudo-stimulation group has 40 patients with dTMS intervention using sham coils (with the same parameters as real dTMS and generating the same noise as real coils, but without the magnetic field). It is given once per day, for 28 days, with a total of 28 treatments.
  Interventions: Device: Sham deep transcranial magnetic stimulation; Other: Basic treatment

INTERVENTIONS:
Device: Deep transcranial magnetic stimulation — Neuronavigation: The coil is positioned 4cm in front of the scalp point and foot motor cortex, corresponding to the ACC. The Brainways H7 coil with fluid cooling is used to obtain a greater depth of stimulation, up to about 6 cm below the cortex.
  dTMS intervention: The intervention targets are at the left and right ACC, once per day, for 28 days. A total of 28 treatments are given. Stimulation mode: stimulation frequency 1Hz, stimulation intensity 100% RMT, number of pulses 150, sequence interval 20s, total 6 trials, 900 pulses.
  Arms: dTMS treatment group
Device: Sham deep transcranial magnetic stimulation — Neuronavigation: The sham coil is positioned 4 cm in front of the scalp point and foot motor cortex, corresponding to the ACC.
  Sham dTMS intervention: The intervention targets are at the left and right ACC (The sham coil has the same parameters as real dTMS and generating the same noise as real coils, but without the magnetic field), once per day, for 28 days. A total of 28 treatments are given.
  Arms: pseudo-stimulation group
Other: Basic treatment — According to national and international guidelines for the treatment of eating disorders, the basic treatment for patients is nutritional therapy, that is, regular and quantitative dietary treatment, with three regular meals followed by a snack meal 2 hours after the regular meal. Both groups received the same nutritional treatment.

SUMMARY:
Hypothesis of "AN-ACC pathological network" suggests that ACC overactivation and abnormal functional connectivity with other brain regions is the neuropathological mechanism for the onset of AN. Currently, rare studies have been conducted on dTMS targeting ACC as an intervention in patients with AN. In this research, dTMS, a neuroregulatory technology, is used for the first time to intervene with ACC in the treatment of adult AN. A randomized controlled study design is adopted, in which patients with AN are divided into the dTMS treatment group and the pseudo-stimulation group by 1:1 randomization, followed by 6-week intervention and half-year follow up, to clarify the near-term and long-term efficacy and safety of the dTMS treatment. Meanwhile, baseline fMRI data will be extracted and combined with clinical features to establish an efficacy prediction model, which will provide theoretical and practical basis for the pioneering ACC-targeted dTMS treatment in China, helping to establish a new type of intervention program for AN, with expected results of innovation.

DETAILED DESCRIPTION:
Building on the previous foundation and literature review, we found that ACC is closely related to the core symptoms of AN, and proposed the hypothesis of "AN-ACC pathological network", suggesting that ACC overactivation and abnormal functional connectivity with other brain regions (anterior frontal lobe, parietal lobe, precuneus, and striatum) is the neuropathological mechanism for the onset of AN.

Currently, rare studies have been conducted on dTMS targeting ACC as an intervention in patients with AN. In this research, dTMS, a neuroregulatory technology, is used for the first time to intervene with ACC in the treatment of adult AN. A randomized controlled study design is adopted, in which patients with AN are divided into the dTMS treatment group and the pseudo-stimulation group by 1:1 randomization, followed by a 28-day intervention (once a day) and half-year follow up, to clarify the near-term and long-term efficacy and safety of the dTMS treatment. Patients in both groups undergo fMRI examinations, complete delay discounting task (DDT) and body image task before and after each treatment session. Efficacy is judged by a weight gain of 4 kg in the four weeks following the intervention. Symptoms, psychometrics and side effect questionnaires are followed up at baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 ( after completion of treatment).

Meanwhile, baseline fMRI data will be extracted and combined with clinical features to establish an efficacy prediction model. We will explore factors predictive of dTMS efficacy in AN patients of dTMS treatment group, divided into two groups according to whether dTMS is effective or not after treatment (defined as a weight gain of 4 kg in the four weeks following the intervention), using pre-treatment (baseline) demographic information, psychological assessment questionnaires, and neuroimaging data in the two groups. This will provide theoretical and practical basis for the pioneering ACC-targeted dTMS treatment in China, helping to establish a new type of intervention program for AN, with expected results of innovation.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-35 years, right handedness.
* Above primary education.
* Meet the diagnostic criteria of AN in DSM-V, and13.0 kg/m2 ≤ body mass index (BMI)<18.5 kg/m2.
* No systemic nutritional therapy, psychiatric medication or any form of psychotherapy have been received within 1 month before enrollment.
* Able to understand the nature of this study and sign an informed consent form.

Exclusion Criteria:

* Diagnosed with a DSM-5 disease other than anorexia nervosa, or at high risk of suicide, strong impulsive behavior as well as anti-social behavior.
* With severe physical or cognitive impairment.
* Not able to undergo MRI.
* Considered unsuitable for enrollment in this clinical trial for other reasons.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI). | whin 4 weeks after completion of treatment
  Calculation: BMI = weight (kg) divided by the square of height (m)

SECONDARY OUTCOMES:
1.Eating Disorder Examination Questionnaire (EDE-Q6.0) | baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 ( after completion of treatment).
  Eating Disorder Examination Questionnaire can assess the core symptoms of eating disorders, including behavioral and psychological characteristics, and rate their frequency and intensity, which can assess the severity of the eating disorder. It consists of 4 subscales, including dietary restriction, eating concerns, body image concerns, and weight concerns.
2.Eating Disorder Inventory (EDI-II) | baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 ( after completion of treatment).
  It is a commonly used scale for assessing cognitive-behavioral symptoms of eating disorders and is used to assess the severity of eating disorders. The scale contains 91 items divided into 8 subscales and 3 temporary subscales, including the pursuit of thinness, bulimia, body dissatisfaction, feelings of ineffectiveness, perfectionism, mistrust of others, introspection, maturity fears, abstinence, impulsive regulation and social insecurity.
3.Beck Depression Inventory (BDI) | baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 ( after completion of treatment).
  The BDI consists of 21 items and assesses the patient's accompanying feelings of depression over the past 2 weeks.
4.Beck Anxiety Inventory (BAI) | baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 ( after completion of treatment).
  The BAI consists of 21 items and assesses the patient's accompanying feelings of anxiety over the past 1 week.
5. Self-assessed Compulsive Questionnaire for Eating Disorders (SR-YBC-EDS) | baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 ( after completion of treatment).
  The SR-YBC-EDS was developed based on the Yale-Brown Compulsive Questionnaire for Eating Disorders (YBC-EDS), consisting of two parts: the first part is a list of 65 symptomatic items, which is used to identify the subjects' obsessive-compulsive symptoms, and the second part is a list of 8 core items, which is used to assess the frequency and severity of obsessive-compulsive symptoms. All parts contain two dimensions: preoccupation and ritual behavior.
6. Body Image Tasks | baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 (after completion of treatment).
  Tasks that address excessive concerns about body shape/weight include the following two parts:
  Body size estimation: The screen will present the above 30 body size pictures sequentially, the subjects will view the body size pictures in 4000ms, and then evaluate the body size of the body pictures in 4000ms, with a score of 1 representing "very low body weight", 4 representing "very overweight", and 4 representing "very overweight". A score of 1 represents "very low weight" and a score of 4 represents "very overweight".
  Body compare task: The screen will present the above 30 body images in turn, the subjects will have 4000ms to view their own images (with randomized distortions), and then they will have 4000ms to compare their actual body shape with the body shape in the images and assess their emotional level. 1 point represents "very calm" and 4 for "very anxious".
7. Delay Discounting Task (DDT task) | baseline, day 28 (at the end of treatment), and weeks 4, 8, 12 and 24 (after completion of treatment).
  The study uses a DDT task in a food choice scenario to assess inhibitory impulses. The task requires subjects to make a decision between choosing a small reward in the present or a large reward in the future. Inhibition to choose a small reward in the present implies a strong intertemporal decision-making ability. The task begins with an assessment of their hunger, willingness to eat, and emotional feelings at the moment. Then they are asked to rate 40 pictures of food on a scale of 0 to 10 on five dimensions: familiarity, craving, positive and negative emotions, emotional intensity, and eating control. Pictures of foods with craving scores >7 and eating control <5, as well as matched in familiarity and emotion for use in the ensuing delay discounting task. The choice is made by pressing a button: Patients choosing to get less food immediately are given fewer coupons after the delay. But those waiting for a period of time to get more food are given more coupons after the delay.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Chen, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Jue Chen, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and baseline characteristics of participants.
Supporting Information: Study Protocol, SAP
Time Frame: Researchers will share data when the study is completed in December 2026.
Access Criteria: dTMS; anorexia nervosa; anterior cingulate cortex

REFERENCES:
- [Background] Kodama N, Moriguchi Y, Takeda A, Maeda M, Ando T, Kikuchi H, Gondo M, Adachi H, Komaki G. Neural correlates of body comparison and weight estimation in weight-recovered anorexia nervosa: a functional magnetic resonance imaging study. Biopsychosoc Med. 2018 Oct 31;12:15. doi: 10.1186/s13030-018-0134-z. eCollection 2018. PMID 30450124
- [Background] King JA, Bernardoni F, Geisler D, Ritschel F, Doose A, Pauligk S, Pasztor K, Weidner K, Roessner V, Smolka MN, Ehrlich S. Intact value-based decision-making during intertemporal choice in women with remitted anorexia nervosa? An fMRI study. J Psychiatry Neurosci. 2020 Mar 1;45(2):108-116. doi: 10.1503/jpn.180252. PMID 31595737
- [Background] Yuan S, Wu H, Wu Y, Xu H, Yu J, Zhong Y, Zhang N, Li J, Xu Q, Wang C. Neural Effects of Cognitive Behavioral Therapy in Psychiatric Disorders: A Systematic Review and Activation Likelihood Estimation Meta-Analysis. Front Psychol. 2022 May 3;13:853804. doi: 10.3389/fpsyg.2022.853804. eCollection 2022. PMID 35592157
- [Background] Bersani FS, Minichino A, Enticott PG, Mazzarini L, Khan N, Antonacci G, Raccah RN, Salviati M, Delle Chiaie R, Bersani G, Fitzgerald PB, Biondi M. Deep transcranial magnetic stimulation as a treatment for psychiatric disorders: a comprehensive review. Eur Psychiatry. 2013 Jan;28(1):30-9. doi: 10.1016/j.eurpsy.2012.02.006. Epub 2012 May 3. PMID 22559998
- [Background] Roth Y, Tendler A, Arikan MK, Vidrine R, Kent D, Muir O, MacMillan C, Casuto L, Grammer G, Sauve W, Tolin K, Harvey S, Borst M, Rifkin R, Sheth M, Cornejo B, Rodriguez R, Shakir S, Porter T, Kim D, Peterson B, Swofford J, Roe B, Sinclair R, Harmelech T, Zangen A. Real-world efficacy of deep TMS for obsessive-compulsive disorder: Post-marketing data collected from twenty-two clinical sites. J Psychiatr Res. 2021 May;137:667-672. doi: 10.1016/j.jpsychires.2020.11.009. Epub 2020 Nov 4. PMID 33183769
- [Background] Carmi L, Alyagon U, Barnea-Ygael N, Zohar J, Dar R, Zangen A. Clinical and electrophysiological outcomes of deep TMS over the medial prefrontal and anterior cingulate cortices in OCD patients. Brain Stimul. 2018 Jan-Feb;11(1):158-165. doi: 10.1016/j.brs.2017.09.004. Epub 2017 Sep 6. PMID 28927961
- [Background] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199
- [Background] Lipsman N, Lam E, Volpini M, Sutandar K, Twose R, Giacobbe P, Sodums DJ, Smith GS, Woodside DB, Lozano AM. Deep brain stimulation of the subcallosal cingulate for treatment-refractory anorexia nervosa: 1 year follow-up of an open-label trial. Lancet Psychiatry. 2017 Apr;4(4):285-294. doi: 10.1016/S2215-0366(17)30076-7. Epub 2017 Feb 24. PMID 28238701
- [Background] Karaszewska D, Cleintuar P, Oudijn M, Lok A, van Elburg A, Denys D, Mocking R. Efficacy and safety of deep brain stimulation for treatment-refractory anorexia nervosa: a systematic review and meta-analysis. Transl Psychiatry. 2022 Aug 15;12(1):333. doi: 10.1038/s41398-022-02102-w. PMID 35970847